CLINICAL TRIAL: NCT06277960
Title: A Prospective, Single-center, Single-arm Clinical Study to Evaluate the Safety and Effectiveness of Percutaneous Intramyocardial Septal Radiofrequency Ablation System in the Treatment of Hypertrophic Obstructive Cardiomyopathy
Brief Title: Septal Ablation for Obstructive HCM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SuZhou Sinus Medical Technologies Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNS2301
Record Dates: First submitted 2024-01-27; First posted 2024-02-26 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Hypertrophic Obstructive Cardiomyopathy (HOCM)
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- percutaneous intramyocardial septal radiofrequency ablation system (Experimental)
  Interventions: Device: percutaneous intramyocardial septal radiofrequency ablation system

INTERVENTIONS:
Device: percutaneous intramyocardial septal radiofrequency ablation system — The device is introduced into the right ventricle and performs ablation treatment on the hypertrophic interventricular septum.

SUMMARY:
Hypertrophic cardiomyopathy (HCM) is a common clinical genetic-related disease, with a global incidence of 0.2%-0.5%, but only a few cases (10-20%) have been clinically diagnosed. About 70% of them are hypertrophic obstructive cardiomyopathy (HOCM), these HOCM patients have significant clinical symptoms, including progressively increasing fatigue, angina, exertional dyspnea, and syncope. Conservative medications are used to treat the vast majority of patients. Invasive therapy, which includes surgical myectomy, percutaneous transluminal septal myocardial ablation(PTSMA), percutaneous intramyocardial septal radiofrequency ablation (PIMSRA) and percutaneous endocardial septal radiofrequency ablation (PESA) is introduced to patients with refractory symptoms or drug resistance. However, surgical operations are complicated and high risk procedures with high mortality. Interventional approaches are very difficult to perform and therefore the application is limited.

Previous researches have shown that interventricular septal radiofrequency ablation could effectively reduce the left ventricular outflow tract pressure gradient (LVOTG), thereby treating obstructive hypertrophic cardiomyopathy (HOCM). This device is based on the same radiofrequency ablation energy principle, however, the catheter is introduced into the right ventricle and performs ablation treatment on the hypertrophic interventricular septum, which is potentially a lower risk route of access for septal ablation than currently attempted interventional approaches.

The purpose of this study is to evaluate the safety and efficacy of percutaneous intramyocardial septal ablation catheters in the treatment of obstructive hypertrophic cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old ≤ age ≤ 75 years old, no gender limit.
2. Subject has pressure gradient of left ventricular outflow tract (LVOT) ≥50 mmHg（with Systolic Anterior Motion）in the resting-state or after exercise stress test.
3. Subject with New York Heart Association (NYHA) cardiac function ≥ II grade.
4. Subject with adequate drug treatment is not effective or cannot tolerate side effects of the drug.
5. Subject was informed of the nature of the clinical study and agreed to participate in all the requirements of the clinical study, signed an ethics committee-approved informed consent form before conducting any special examinations and/or treatments related to the clinical study.

Exclusion Criteria:

1. Subject is pregnant, lactating, or planned to conceive during a clinical study.
2. Subject with interventricular septal thickness ≥ 30mm.
3. Subject has undergone other ventricular septal volume reduction surgeries.
4. Subject with complete right bundle branch block on electrocardiogram.
5. Subject with Sudden Cardiac Death Index ≥ 10%.
6. Subject combined with other heart diseases requires surgical treatment.
7. Subject with heart failure(Defined as resting heart failure after intensive anti-heart failure therapy, left ventricular fraction of ejecting< 40%).
8. Subject is mentally incapacitated or unable to understand the study requirements.
9. Subject has participated in other clinical trials within 3 months.
10. The investigator determines that there is any situation that affects the safety of the subjects or interferes with the evaluation of test results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-03-28 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
30-day major adverse clinical events (MACE) | 30-day
  30-day major adverse clinical events (MACE), including death, emergency surgery, severe pericardial effusion bleeding requiring pericardiocentesis or surgery, atrioventricular block, heart perforation, and surgery-related stroke.

SECONDARY OUTCOMES:
Technical success rate | 30-day
  Technical success rate: the radiofrequency ablation catheter reaches the required treatment site, successfully completes the ablation, and is successfully withdrawn from the body.
Short Form 36 (SF-36) health survey questionnaire | 90-day
  The life quality score of SF-36 would significantly improved after the procedure. The higher scores mean a better outcome.
Improvement of left ventricular outflow tract gradient (LVOTG) | 6 months
  The improvement of LVOTG at post-procedure,30 days,3 months and 6 months after procedure. If the pressure gradient is reduced, the symptom will improve.
Improvement of NYHA functional classification | 6 months
  The improvement of NYHA functional class at post-procedure,30 days,3 months and 6 months after procedure. The lower class mean a better outcome.
6-min walk distance | 6 months
  The increase of 6-min walk distance at post-procedure,30 days,3 months and 6 months after procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Shaw Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided